CLINICAL TRIAL: NCT05168956
Title: Apparent Characteristics of Genealogical Representations of Perpetrators of Sexual Violence.
Brief Title: Characteristics of Genealogical Representations of Perpetrators of Sexual Violence.
Acronym: CARG-AVS
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN1052021/CHUSTE
Record Dates: First submitted 2021-12-10; First posted 2021-12-23 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Sexual Offence
Keywords: Sexual abuse; family; sexual offenders; incest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sexual offender: Patients followed up in the sexual offender's department of University Hospital of Saint Etienne will be included.
  Interventions: Other: Collect data of medical record

INTERVENTIONS:
Other: Collect data of medical record — Collect data of medical record:
  * Genealogy characteristics
  * Family characteristics: Number of members in the sibling, rank in the sibling / incestuous relationships or not
  * Graphic representation: age / gender / age at time of sexual assault / whether or not a victim of sexual violence / education / family dynamics / living environment during childhood / Criminal category

SUMMARY:
Two French studies report that 25% of sexual abuse occurs in intrafamily sphere. To be victim of sexual abuse leads to cognitive troubles and redesign of psychological processes. Lot of studies report that offenders had been victims (30-97%). How psychological redesign is destroying genealogical representation and hinders the proper construction of family ties.

This study to study characteristics data about family, and how the patients see it, from medical records of a specific department for sexual offenders in University Hospital of Saint Etienne. Study is realized blind from criminal categories. Data are gathered with a standardized grid, to guarantee reproducibility of data collection.

DETAILED DESCRIPTION:
The CARG-AVS study does not involve any additional examinations or consultations compared to usual practice. It consists of collecting information from patients' medical records.

ELIGIBILITY:
Inclusion Criteria:

* Patients followed up in the sexual offender's department of University Hospital of Saint Etienne.
* Patients who did the nursing assessment at time of analysis.

Exclusion Criteria:

* Patients in the preliminary follow up in the department
* Refusal to participate at this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients followed up in the sexual offender's department of University Hospital of Saint Etienne will be included.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2022-04-05 (Actual); Primary Completion 2022-04-28 (Actual); Study Completion 2022-04-28 (Actual)

PRIMARY OUTCOMES:
Characteristic of family | the day of the medical file review
  Structural characteristic of family tree according to the penal category Collected in medical record.

SECONDARY OUTCOMES:
Family members | the day of the medical file review
  Number of members in the sibling, rank in the sibling collected in medical record.
Incestuous relationships | the day of the medical file review
  Number of incestuous relationships in the family collected in medical record.
Psychological traumatisms: sexual abuse | the day of the medical file review
  Existence of psychological traumatisms: sexual abuse collected in medical record.
Psychological traumatisms: brutal deat | the day of the medical file review
  Existence of psychological traumatisms: brutal deat collected in medical record.
Psychological traumatisms: severe illness | the day of the medical file review
  Existence of psychological traumatisms: severe illness collected in medical record.
Psychological traumatisms: suicide | the day of the medical file review
  Existence of psychological traumatisms: suicide collected in medical record.
Criminal category | the day of the medical file review
  Criminal category collected in medical record.

CONTACTS AND LOCATIONS:
Overall Officials: Tristan GABRIEL, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No